CLINICAL TRIAL: NCT07288190
Title: A Multisite, Open-label, Randomized Crossover Study Comparing Adherence to a Single Daily Dual Prevention Pill (DPP) Versus FTC/TDF and Combined Oral Contraception Separate Pill Dosing (2PR), Given for Pre-exposure Prophylaxis and Pregnancy Prevention in Women
Brief Title: Phase 2b, Open Label, Multisite, Randomized Crossover Study of DPP Versus 2PR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 104; UM1AI068619 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy; HIV Infections
Keywords: Pre-exposure Prophylaxis (PrEP); Contraception; Dual Prevention Pill (DPP); Pregnancy Prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Phase 2b, open label, multisite, randomized crossover study of DPP versus 2PR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DPP/2PR/Choice (Experimental): Daily DPP for 12 weeks followed by daily 2PR for 12 weeks followed by 24 weeks of Choice
  Interventions: Drug: DPP; Drug: 2PR; Drug: Free Choice
- 2PR/DPP/Choice (Experimental): Daily 2PR for 12 weeks followed by daily DPP for 12 weeks followed by 24 weeks of Choice
  Interventions: Drug: DPP; Drug: 2PR; Drug: Free Choice

INTERVENTIONS:
Drug: DPP — Daily, single, co-formulated, FTC/TDF + combined ethinyl estradiol/levonorgestrel oral contraceptive pill
Drug: 2PR — Daily, two-pill regimen of oral FTC/TDF and ethinyl estradiol/levonorgestrel oral contraceptive pill
Drug: Free Choice — Choice of either DPP or 2PR

SUMMARY:
To evaluate adherence to a single dual-prevention pill (DPP) compared with a two-pill regimen (2PR) for pre-exposure prophylaxis (PrEP) and pregnancy prevention in women without HIV.

DETAILED DESCRIPTION:
To evaluate adherence to a single DPP consisting of co-formulated Tenofovir Disoproxil Fumarate and Emtricitabine (FTC/TDF) plus combined ethinyl estradiol/levonorgestrel oral contraceptive (COC), compared with a two-pill regimen (2PR) consisting of daily oral FTC/TDF pill and combined COC pill, for pre-exposure prophylaxis PrEP and pregnancy prevention in women without HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 through 39 years old (inclusive) at Screening.
* Adults must be able and willing to provide informed consent. Adolescents (16- and 17-year-olds) will be consented according to applicable local guidelines, by obtaining participant assent and where applicable parental or guardian permission.
* Able and willing to provide adequate locator information.
* Able and willing to comply with all study procedures.
* Must be post-menarche and pre-menopausal and could potentially become pregnant.
* Sexually active, defined as having had penile-vaginal sex within the 3 months before Screening (per self-report)
* Negative pregnancy test at Screening and Enrollment.
* Does not intend to become pregnant within the next 12 months.
* Willing to use COCs for at least 48 weeks as their method of contraception.
* HIV negative at Screening and Enrollment.
* Willing to use oral PrEP for at least 48 weeks.
* Hepatitis B (HBV) surface antigen (HbsAg) negative per blood test at Screening.
* Hepatitis C (HCV) negative at Screening.
* Normal estimated creatinine clearance (eCrCl) ≥ 60 ml/min per blood test at Screening.

Exclusion Criteria:

* Intolerance, adverse reaction, or laboratory abnormality associated with PrEP use in the past.
* Unable to become pregnant e.g., had a tubal ligation or hysterectomy or otherwise lacks a uterus, or is currently using another form of contraception.
* Medically ineligible for combined hormonal contraception and specifically COCs per World Health Organization (WHO) medical eligibility criteria for contraceptive use or similar local medical eligibility guidelines (e.g., Centers for Disease Control and Prevention eligibility criteria).
* Medically ineligible for PrEP based on WHO and/or local guidelines.
* Using or planning to use another pregnancy prevention product other than oral contraception (condoms are permitted) during the next 48 weeks.
* Using or planning to use another HIV prevention product other than condoms during the next 48 weeks.
* Any other condition the clinician feels would jeopardize the health and wellbeing of the participant

Ages: 16 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women
Enrollment: 300 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
PrEP adherence to DPP during randomized crossover period 1 | Week 12
  Intraerythrocytic Tenofovir Diphosphate (TFV-DP) concentrations in dried blood spot (DBS)
PrEP adherence to 2PR during randomized crossover period 1 | Week 12
  Intraerythrocytic TFV-DP concentrations in DBS
PrEP adherence to DPP during randomized crossover period 2 | Week 24
  Intraerythrocytic TFV-DP concentrations in DBS
PrEP adherence to 2PR during randomized crossover period 2 | Week 24
  Intraerythrocytic TFV-DP concentrations in DBS

SECONDARY OUTCOMES:
PrEP adherence to DPP during Choice period | Week 48
  TFV-DP concentrations in DBS
PrEP adherence to 2PR during Choice period | Week 48
  TFV-DP concentrations in DBS
PrEP adherence to DPP during Choice period | Week 48
  Self-reported adherence
PrEP adherence to 2PR during Choice period | Week 48
  Self-reported adherence
Acceptability of DPP during crossover period | Week 24
  Answers to acceptability questionnaire based on overall acceptability measure as well as a range of acceptability dimensions (e.g., product size, color, dosing, etc.)
Acceptability of 2PR during crossover period | Week 24
  Answers to acceptability questionnaire based on overall acceptability measure as well as a range of acceptability dimensions (e.g., product size, color, dosing, etc.)
Acceptability of DPP during Choice period | Week 48
  Answers to acceptability questionnaire based on overall acceptability measure as well as a range of acceptability dimensions (e.g., product size, color, dosing, etc.)
Acceptability of 2PR during Choice period | Week 48
  Acceptability of 2PR based on answers to acceptability questionnaire based on overall acceptability measure as well as a range of acceptability dimensions (e.g., product size, color, dosing, etc.)
Preference for DPP | Day 0
  Preference of DPP at enrollment
Preference for DPP | Week 24
  Preference of DPP at completion of the crossover phase of the study
Preference for 2PR | Day 0
  Preference of 2PR at enrollment
Preference for 2PR | Week 24
  Preference of 2PR at completion of the crossover phase of the study
PrEP persistence on DPP during the Choice period | Week 48
  Proportion of participants still using their chosen regimen at end of the Choice period
PrEP persistence on 2PR during the Choice period | Week 48
  Proportion of participants still using their chosen regimen at end of the Choice period
Overall tolerability of DPP | Week 48
  Tolerability
Overall tolerability of 2PR | Week 48
  Tolerability
Tolerability of DPP during the crossover period | Week 24
  Tolerability
Tolerability of 2PR during the crossover period | Week 24
  Tolerability
Tolerability of DPP during the Choice period | Week 48
  Tolerability
Tolerability of 2PR during the Choice period | Week 48
  Tolerability
Overall side effects of DPP | Week 48
  Grade 2+ Adverse Events (AE)
Overall side effects of 2PR | Week 48
  Grade 2+ AE
Side effects of DPP during the crossover period | Week 24
  Grade 2+ AE
Side effects of 2PR during the crossover period | Week 24
  Grade 2+ AE
Side effects of DPP during the Choice period | Week 48
  Grade 2+ AE
Side effects of 2PR during the Choice period | Week 48
  Grade 2+ AE
Overall unintended IPV of DPP | Week 48
  Intimate Partner Violence (IPV)
Overall unintended IPV of 2PR | Week48
  IPV
Unintended IPV of DPP during the crossover period | Week 24
  IPV
Unintended IPV of 2PR during the crossover period | Week 24
  IPV
Unintended IPV of DPP during the Choice period | Week 48
  IPV
Unintended IPV of 2PR during the Choice period | Week 48
  IPV
Overall unintended pregnancy of DPP | Week 48
  Pregnancy
Overall unintended pregnancy of 2PR | Week 48
  Pregnancy
Unintended pregnancy of DPP during the crossover period | Week 24
  Pregnancy
Unintended pregnancy of 2PR during the crossover period | Week 24
  Pregnancy
Compare unintended pregnancy of DPP during the Choice period | Week 48
  Pregnancy
Compare unintended pregnancy of 2PR during the Choice period | Week 48
  Pregnancy
Overall unintended HIV incidence of DPP | Week 48
  HIV incidence
Overall unintended HIV incidence of 2PR | Week 48
  HIV incidence
Unintended HIV incidence of DPP during the crossover period | Week 24
  HIV incidence
Unintended HIV incidence of 2PR during the crossover period | Week 24
  HIV incidence
Unintended HIV incidence of DPP during the Choice period | Week 48
  HIV incidence
Unintended HIV incidence of 2PR during the Choice period | Week 48
  HIV incidence

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, Study Chair — Population Council; Harriet Nuwagaba-Biribonwoha, MD, Study Chair — ICAP at Columbia University

IPD SHARING:
Plan to Share IPD: Yes
For studies within two years of primary objective(s) publication, de-identified individual participant data that underlie results in a publication will be provided upon request. For studies more than two years from the primary objective(s) publication, de-identified datasets will be available upon request (Public Use Datasets).
Supporting Information: Study Protocol, SAP
Time Frame: Investigators may request de-identified datasets in order to duplicate published results, as required by specific journals. Otherwise, de-identified datasets will be made available upon request, two years following publication of the primary results manuscript.
Access Criteria: Researchers aiming to duplicate published results or who provide a methodologically sound proposal for use of the data may submit a request for access to data that has informed published results by sending an email to HPTN-Data-Access@scharp.org. To access available de-identified datasets, investigators must complete the request form on the Atlas website. Researchers of approved requests will need to sign an HIV Prevention Trials Network (HPTN) Data Use Agreement before receiving the data and agree to use the provided acknowledgement statement.